CLINICAL TRIAL: NCT05489536
Title: A Web/Smartphone-based Lifestyle Program for the Prevention of Gestational Diabetes Mellitus (GDM) in Malaysia: Optimizing Gestational Weight Gain (GWG)
Brief Title: Optimizing Gestational Weight Gain for Prevention of Gestational Diabetes Mellitus in Malaysia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: The World Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Chan Yoke Mun, Professor, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPM19062022
Record Dates: First submitted 2022-07-06; First posted 2022-08-05 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Pregnant Women
Keywords: Health and Nutrition Education (HNE) Resources; Web/smartphone-based Lifestyle Program; Gestational Diabetes Mellitus; Gestational Weight Gain
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Web/smartphone-based Lifestyle Program Intervention Group (Experimental): As this study is designed specifically to isolate the effect of introducing the web/app into the existing care pathway, the intervention group will receive standard prenatal care provided by health clinics and the web/smartphone app.
  Interventions: Behavioral: A web/smartphone-based lifestyle program package
- Control Group (No Intervention): A standard usual prenatal care includes ten clinic visits for routine pregnancy checks (weight gain, iron status, blood pressure, fasting blood glucose etc.)

INTERVENTIONS:
Behavioral: A web/smartphone-based lifestyle program package — There are two platforms for the lifestyle program, namely Health and Nutrition Education (HNE) website and HNE app. The participants are requested to download and register on the HNE website and the HNE app. The HNE app is Android and IOS compatible. Both the HNE website and app are designed to support self-directed learning and independently monitor their GWG and dietary intake during pregnancy. Both the HNE website and app will be passcode protected throughout the study period such that access is restricted to only participants in the intervention group.
  The web/smartphone-based lifestyle program package consists of:
  I. Health and Nutrition Education (HNE) resources II. Gestational Weight Gain (GWG) monitoring III. Dietary intake monitoring
  Arms: A Web/smartphone-based Lifestyle Program Intervention Group

SUMMARY:
Gestational weight gain (GWG) has been closely related to health outcomes, particularly in gestational diabetes mellitus (GDM). Pregnant women may be particularly motivated to make healthy lifestyle changes. Previous studies showed that lifestyle modification interventions (diet and exercise) may be successful in reducing GWG in high-risk women but their effects on the incidence of GDM and other adverse perinatal outcomes have been limited. The research question for the future full randomized trial is whether an optimizing healthy GWG programme focusing on lifestyle (diet and physical activity) feasible to decrease the risk of GDM in a developing country. Thus, this study aims to evaluate the effectiveness of a web/smartphone-based lifestyle program in optimizing gestational weight gain (GWG) to prevent the incidence of GDM.

DETAILED DESCRIPTION:
General objective: To determine the effectiveness of a web/smartphone-based lifestyle program on optimizing gestational weight gain (GWG) to prevent the incidence of GDM.

Specific objectives:

1. To compare changes in the primary outcome (incidence of GDM) between pregnant mothers receiving web/smartphone-based lifestyle program (i.e. intervention group) and pregnant mothers not receiving web/smartphone-based lifestyle program (i.e. control group).
2. To compare changes in the secondary outcomes (GWG, dietary intake and physical activity) between pregnant mothers receiving web/smartphone-based lifestyle program (i.e. intervention group) and pregnant mothers not receiving web/smartphone-based lifestyle program (i.e. control group).

Study location: A total of nine (9) states are randomly selected to represent the Northern, Southern, East Coast and central regions of Peninsular Malaysia. The states are then randomly assigned to either the intervention states or control states. All maternal and child health (MCH) clinics in the top five highest populated districts are purposively selected.

Study design: This is a cluster-randomized, controlled trial (RCT), whereby states as clusters and will be randomly allocated into either intervention or control group. All pregnant women in each cluster will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian women
* At any trimester of pregnancy
* All ethnicities (Malays, Chinese or Indians)
* With or without diseases (diabetes mellitus with/ without insulin, hypertension, dyslipidaemia, overweight/ obese)

Exclusion Criteria:

* Medical diagnosis with major psychiatric problems (bipolar depression, schizophrenia, suicidal risk)
* Severe comorbidities (eg cardiac diseases, kidney diseases severe anemia) that require specific interventions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20000 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of GDM | 9 months after pregnancy
  All pregnant women who attend MCH clinics for prenatal checkups are required to take a standardized 2-hour 75g Oral Glucose Tolerance Test (OGTT) between 28 - 32nd weeks of gestation. Women are requested to report their fasting plasma glucose (FPG) level and 2-hour plasma glucose (2hPG) level. Gestational diabetes mellitus (GDM) is defined as either one or both FPG ≥ 5.1 mmol/L or 2hPG ≥ 7.8 mmol/L. The percentage of women with GDM in both intervention and control groups will be calculated.

SECONDARY OUTCOMES:
Gestational Weight Gain | 9 months after pregnancy
  Women are requested to report their pre-pregnancy weight, the measured height at the maternal and child health (MCH) clinic, as well as the weight at each trimester. If the women could not remember their pre-pregnancy weight, the weight at early pregnancy will be used to estimate pre-pregnancy body mass index (BMI). Total GWG is defined as the last measured weight in the third trimester minus the pre-pregnancy weight or early pregnancy weight, referring to the Institute of Medicine (IOM, 2009). The rate of GWG in the second and third trimesters is defined as the average weekly weight gain in that trimester. Total GWG and rate of GWG will be then categorized as inadequate, adequate or excessive for each category of pre-pregnancy BMI. Percentage of women with insufficient, normal and excessive weight gain will be calculated. The differences in GWG between intervention and control groups will be compared.
Dietary Intake | 9 months after pregnancy
  Dietary intake of women at each trimester will be assessed through a semi-quantitative food frequency questionnaire (sFFQ). Women are asked about the frequency and amount (serving size) of intake of each food item. Daily energy, nutrients intake and number of servings (grams) for each food group will be calculated. The differences in dietary intake between intervention and control groups will be compared.
Physical Activity | 9 months after pregnancy
  Pregnancy Physical Activity Questionnaire (PPAQ) will be used to determine the physical activity level of pregnant women at each trimester. The PPAQ is a semi-quantitative questionnaire that requests respondents to report the time spent participating in 30 activities, including household/caregiving (12 activities), occupational (5 activities), sports/exercise (7 activities), transportation (3 activities), and sedentary (3 activities). Total activity will be calculated as the sum of all intensity activities and type scores. The differences in physical activity between intervention and control groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Zalilah Mohd Shariff, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (9):
- Malaysia (9):
  - Health Clinics in Southern of Peninsular Malaysia, Johor Bahru, Johor
  - Health Clinics in Northern of Peninsular Malaysia, Alor Star, Kedah
  - Health Clinics in East Coast of Peninsular Malaysia, Kota Bharu, Kelantan
  - Health Clinics in Southern of Peninsular Malaysia, Malacca, Malacca
  - Health Clinics in Southern of Peninsular Malaysia, Seremban, Negeri Sembilan
  - Health Clinics in Central of Peninsular Malaysia, Ipoh, Perak
  - Health Clinics in Northern of Peninsular Malaysia, George Town, Pulau Pinang
  - Health Clinics in Central of Peninsular Malaysia, Petaling Jaya, Selangor
  - Health Clinics in East Coast of Peninsular Malaysia, Kuala Terengganu, Terengganu

IPD SHARING:
Plan to Share IPD: No